CLINICAL TRIAL: NCT04664127
Title: Clinical and Immunological Study of the Efficacy and Safety of Combined Treatment of Patients With Severe Herpes Simplex (HSV) Infection) by Acyclic Nucleoside Valacyclovir and Interferon Inducer Kagocel
Brief Title: Study of the Efficacy and Safety of Combined Treatment of Patients With Severe Herpes Simplex (HSV) Infection by Valacyclovir and Interferon Inducer Kagocel
Status: Completed | Type: Observational
Sponsor: Nearmedic Plus LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: version 1.0 from 20.10.2017
Record Dates: First submitted 2020-11-27; First posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2019-01

CONDITIONS: Herpes; Herpes Simplex; Herpes Oral; Herpes Simplex 2; Herpes Genitalis
Keywords: herpes simplex; HSV1; HSV2; Herpes Genitalis; Herpes Oral; herpes simplex viruses; Valaciclovir
MeSH Terms: conditions — Herpes Simplex; Herpes Genitalis | interventions — Valacyclovir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Combination therapy (Kagocel + Valacyclovir: n=25): Therapy according to routine practice (including Kagocel). Groups will be splitted during the final data analysis.
  Interventions: Drug: Kagocel+Valacyclovir
- Monotherapy by Valacyclovir (n=20): Therapy according to routine practice. Groups will be splitted during the final data analysis.
  Interventions: Drug: Valacyclovir

INTERVENTIONS:
Drug: Kagocel+Valacyclovir — Group 1-patients with simple severe herpes (HSV-infection orolabial and / or genital localization) treatment [Valacyclovir + Kagocel ° ] (n= 25).
  Treatment: Valacyclovir, 1000 mg orally (2 tablets of 500 mg): 1 time per day for at least 4 months continuously (the rate of suppressive therapy). * Kagocel®, 24 mg orally (2 tablets of 12 mg): 3 times per day, 5 days continuously.
  * - During the study the minimum duration of Valacyclovir suppressive therapy in instruction for medical use that drag was changed from 4 (what was using in our reserch) to 6 months, and the optimal duration of continuous antiviral therapy with PG was changed from 6 to 12 months
  Groups: Combination therapy (Kagocel + Valacyclovir: n=25)
Drug: Valacyclovir — Group 2 -patients with simple severe herpes (HSV-infection orolabial and/or genital localization) receiving treatment [Valacyclovir] (n= 20).
  Scheme of treatment: Valacyclovir, 1000 mg orally (2 tablets of 500 mg): 1 time per day for at least 4 months continuously (a course of suppressive therapy)*.
  * - During the study the minimum duration of Valacyclovir suppressive therapy in instruction for medical use that drag was changed from 4 (what was using in our reserch) to 6 months, and the optimal duration of continuous antiviral therapy with PG was changed from 6 to 12 months.
  Groups: Monotherapy by Valacyclovir (n=20)

SUMMARY:
This study examined the efficacy, safety and benefits of modern treatment and changes in the dynamics of the life of adult patients quality with severe herpes simplex in the current medical practice when combined therapy by acyclic nucleoside Valacyclovir and antiviral agent Kagocel versus monotherapy by Valacyclovir. This study also evaluated the structure of herpesvirus infections and the rate of mixed variants of the course, the rate of exacerbations of herpes simplex, the time of disappearance of human herpesvirus isolation and the features of the immune phenotype of patients taking different types of therapy.

DETAILED DESCRIPTION:
This study was a comparative post-registration prospective non-interventional (observational) scientific study.

This research did not include any procedures or medical interventions except those recommended in the local clinical guidelines and international standards of care. All procedures and evaluations were performed in accordance with routine clinical practice adopted in the Russian Federation and the instructions for the medical use of drugs that patients received.

The following data was collected and analyzed after the end of treatment:

* demography
* disease severity (mild, moderate, severe, continuous relapses)
* data of anamnesis (hereditary and family anamnesis, duration of herpes simplex disease, previous illnesses, duration of treatment, previous treatment of herpes simplex and its efficacy, allergic anamnesis, epidemiological anamnesis, rate and duration of herpes relapses over the past year (with indication of the location of herpes simplex rashes), main diagnosis and complications, ICD-10 code, date and time of the last exacerbation, causes of exacerbation)
* verification of inclusion criteria
* verification of non-inclusion criteria
* prescribed therapy (trade name and prescription scheme, rate, method of administration)
* laboratory tests (4 timelines: 1 - first 6-48 hours; 2 - 6 days after starting of therapy; 3 - 30 days; 4 - 4 months): clinical and biochemical blood tests; serological diagnostics with determination of herpes virus infections's markers: IgM, IgG-HSV1, HSV2; hospital screening of venous blood: anti - HIV-1,2; anti-HCV-total, HBsAg, CSR; microbiological seeding from the tonsils, posterior pharyngeal wall with determination of drug sensitivity; PCR of blood, saliva and/or rash elements; immune status by laser flow cytometry: CD3+, CD4+, CD8+, CD4+/CD8+, CD16+, CD19+; serum immunoglobulins: IgA, IgM, IgG, IgE total.
* medical anamnesis (4 timelines: 1 - first 6-48 hours; 2 - 6 days after starting of therapy; 3 - 30 days; 4 - 4 months) or clinical efficacy: the presence and rate of exacerbations of the disease orolabial, genital and other sites; local complaints; the rate of occurrence of and general symptoms; the rate of epithelialization of the rash's morphological elements; duration of recurrence of the herpes simplex virus and speed of onset of epithelialization; the rate of relapses and exacerbations of herpes simplex on the background of suppressive therapy
* taking other drugs during the study (trade name, prescription scheme)
* compliance with the drugs regimen
* timelines: data of signing the informed consent, start date of the study, date of each patient visit, end date of the study, start date and end date of the taking medicines, duration of patient follow-up)
* quality of life assessment at the end of the study (excellent / good / satisfactory / has not changed)
* adverse events (yes/no, data description)

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old
* The absence of systemic etiotropic antiviral and immunosuppressive therapy for at least a year at the time of inclusion in this study
* Severe herpes simplex (HSV infection with orolabial and / or genital localization) with a recurrence rate of 6 or more for last 12 months.
* The first 6-48 hours after the exacerbation of herpes simplex.
* The following diseases and conditions are missing, usually requiring combination therapy by more than 2 drugs: ophthalmic herpes, visceral herpes, herpetic encephalitis, Kaposi's herpetiform eczema, primary immunodeficiency (PID criteria are given below*), tuberculosis, ARVI and influenza symptoms (not related to herpesviruses), diabetes mellitus, hepatitis B and/or C, autoimmune diseases, HIV infection, other diseases requiring specific treatment (syphilis, gonorrhea), septic conditions, cancer (except of benign skin growths), mental illness, alcohol and/or drug addiction, artificial radiation and/or radiation therapy.
* Standard Valacyclovir therapy prescribed by doctor, or combination therapy by Valacyclovir and Kagocel.

Exclusion Criteria:

* Basic cytostatic therapy, taking systemic glucocorticoids for life indications. Treatment by immunoglobulins and any vaccines for 30 days prior to inclusion in the study.
* Early period (up to 1 month) after any vaccination.
* Pregnancy, including pregnancy planning for 3 months and lactation.
* The presence of a genetic disease or verified primary immunodeficiency.
* Anamnesis of transplantation of organs and tissues.
* Plasmapheresis and blood donation for less than 6 months before the present study.
* Severe kidney and liver damage.
* Any other diseases or conditions that, by the opinion of the researcher, may interfere the patient from being included in the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult men and women with signs of severe herpes simplex.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2018-10-29 (Actual); Study Completion 2018-10-29 (Actual)

PRIMARY OUTCOMES:
Change of the patients proportion with different localizations of herpes simplex exacerbations. | 2 points: before and 6 months after the start of therapy
Change of the rate of exacerbations of orolabial, genital and other localization herpes simplex | 2 points: before and 6 months after the start of antiviral therapy
Change of the number of patients with varying degrees of severity illness | 2 points: before and 6 months after the start of therapy
Change in the number of local complaints (pain, itching, burning, rash) against the background of a recurrence of herpes simplex | up to 6 months

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events (AE) with regards to type and severity of AE (mild, moderate, severe; according to physician's opinion) | up to 6 (12) mounts
Change of the duration of each herpes simplex relapse and the rate of epithelialization | 2 points: before and 6 days after the start of therapy
Change of the occurrence rate of morphological elements of the rash and General symptoms | 4 points: 1-before the start of therapy, 2-6 days after the start of therapy, 3-30 days, 4-4 months
Change of the rate of herpes simplex rash (relapses) | 4 points: 1 - before the start of therapy, 2 - 6 days after the start of therapy, 3 - 30 days, 4 - 4 months
Change of the intensity of herpes simplex exacerbations in points | 4 points: 1-before the start of therapy, 2-6 days after the start of therapy, 3-30 days, 4-4 months
  Herpes simplex exacerbation were local symptoms (according to the patient's assessment: pain, itching, burning, rash); localization of the rash (according to the doctor's assessment: orolabial, genital, other); morphology of the rash (ulcer and / or erosion, vesicle, crust, spot); intensity of the rash (single element, several elements, multiple rashes); enlarged lymph nodes; general symptoms (weakness, drowsiness, decreased physical activity, increased body temperature).
  There was used subjective assessment: 1 point - min, 10 points - max intensity.
Change in the number of herpes viruses in saliva and blood by PCR | 4 points: 1-before the start of therapy, 2-6 days after the start of therapy, 3-30 days, 4-4 months
  Identification of herpes viruses type 1 and 2 (HSV1, HSV2), cytomegalovirus (CMV), Epstein-Barr virus (EBV), herpesvirus type 6 (HHV6, HHV7, HHV8) and assessment of the duration of their isolation.
Change of antibodies titers to herpes simplex viruses type 1 and 2 | 2 points: before the start of therapy and on the 30th day after the start of therapy
  Detection of specific antibodies levels against herpes simplex virus (anti-HSV-1,2 IgM, anti-HSV-1,2 IgG) using ELISA in both groups
Change of immune status parameters (flow cytometry) | 2 points: before treatment and at 30 days after initiation of therapy
  Determination of changes of serum immunoglobulin levels by laser flow cytometry (g / l, UL): IgA, IgM, IgG, IgE total
Change of immune status parameters (flow cytometry) | 2 points: before treatment and at 30 days after initiation of therapy
  Detection of changes of immune status parameters by laser flow cytometry (%): CD3+, CD4+, CD8+, CD4+/CD8+, CD16+, CD19+
Change of lymph nodes sizes (submandibular, axillary, inguinal) according to ultrasound data | 2 points: before and 6 months after the start of therapy
The assessment of quality of life according to questionnaire | up to 6 months after initiation of therapy
  Criteria for evaluating the "Quality of life" indicator were:
  "excellent" - rashes and relapses of herpes simplex (HSV) are absent, physical and mental activity are above average, "good" - rare rashes of HSV (no more than 1-2 times per year), physical and mental activity are average, "satisfactory" - the rash of HSV were less likely (up to 3-4 times per year), physical and mental activity are below average, "has not changed" - the recurrence rate HSV for 6-12 months was same (as before the start of therapy and participation in the study), physical and mental activity are unsatisfactory.

CONTACTS AND LOCATIONS:
Overall Officials: Georgy Vikulov, Ph.D, Principal Investigator — Scientific Information Center for Prevention and Treatment of Viral Infections
Locations (1):
- Scientific Information Center for Prevention and Treatment of Viral Infections, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Vikulov G., Voznesenskiy S. Сombination antiviral therapy of herpes simplex // Vrach. - 2019; 30 (5): 27-34. https://doi.org/10.29296/25877305-2019- 05-05 — http://vrachjournal.ru/25877305-2019-05-05
- See also: Vikulov G.Kh., Voznesenskiy S.L. Combination antiviral therapy in patients with severe herpes simplex virus infections: clinical and immunological characteristics and assessment of patients' quality of life. Infectious diseases. 2019; 17(4): 79-91 — https://www.phdynasty.ru/en/catalog/magazines/infectious-diseases/2019/volume-17-issue-4/37443